CLINICAL TRIAL: NCT03039426
Title: A Randomized Comparison of Bupivacaine Peritoneal and Subcutaneous Infiltration Versus Diclofenac Intramuscular Injection for Postoperative Pain Relief in Patient Undergoing Cesarean Delivery
Brief Title: Postoperative Cesarean Delivery Pain Relief; Diclofenac Versus Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RJBUPI
Record Dates: First submitted 2016-09-28; First posted 2017-02-01 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2017-10

CONDITIONS: Cesarean Delivery
MeSH Terms: interventions — Bupivacaine; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Bupivacaine (Experimental): 0.5% bupivacaine 20ml divided in two; 10 ml intraperitoneal infiltration and 10 ml subcutaneous infiltration
  Interventions: Drug: Bupivacaine
- Group Diclofenac (Active Comparator): diclofenac 75 mg intramuscular, 2 hours postoperation
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Bupivacaine — 0.5% bupivacaine 20ml divided in two; 10 ml intraperitoneal infiltration and 10 ml subcutaneous infiltration
  Arms: Group Bupivacaine
Drug: Diclofenac — diclofenac 75 mg intramuscular, 2 hours postoperation
  Arms: Group Diclofenac

SUMMARY:
This randomized controlled trial, compared postoperative pain score in patient undergoing cesarean delivery between bupivacaine peritoneal and subcutaneous infiltration and diclofenac intramuscular injection

DETAILED DESCRIPTION:
Postoperative cesarean delivery was painful that can effect daily activity, resulted in poor quality of life and required morphine injection to relief pain which had both maternal and breastfeeding infancy side effect. So this study compare efficacy of diclofenac and bupivacaine by measured the pain score and requirement of morphine injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo elective or urgency cesarean delivery at Rajavithi Hospital in 2016-2017

  * Urgency conditions: CPD, fail induction of labor, antepartum hemorrhage without hypovolemic shock, dystocia, previous cesarean section and active labor, malpresentation in labor, macrosomic presentation in labor
* Pregnant women more than 20 years of age
* Gestational age more than 37 week
* Cesarean section under regional or general anesthesia
* Ability to communicating, writing and reading Thai language

Exclusion Criteria:

* Inability to communicating or writing or reading Thai language
* Contraindicated to bupivacaine or diclofenac or morphine
* Pregnant women with emergency conditions
* Have one or more complication of pregnancy
* Intraoperative arrhythmia
* Pregnant women less than 20 years of age
* Regional anesthesia with morphine

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Compared pain score change from baseline at 2, 6 and 24 hours at post-operation between 2 groups by visual analogue scale | 2, 6 and 24 hours post-operation
Compared rescued dose of morphine injection | Within 24 hours post-operation

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Natthida Mekwongtrakarn, Bangkok
  - Rajavithi Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No